CLINICAL TRIAL: NCT07069933
Title: "Repurposing Itraconazole as an Adjuvant Therapy in Treatment of Patients With Acute Myeloid Leukemia: Is it a Hopeful Avenue for Enhancing Treatment Options?"
Brief Title: Repurposing Itraconazole as an Adjuvant Therapy in Treatment of Patients With Acute Myeloid Leukemia: Is it a Hopeful Avenue for Enhancing Treatment Options?
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Noha Mansour, Lecturer of Clinical Pharmacy and Pharmacy Practice, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024-42-2024-120
Record Dates: First submitted 2025-02-14; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control arm (Other): Standard Care
  Interventions: Drug: Chemotherapy
- Interventional arm (Active Comparator): Standard Care plus itraconazole
  Interventions: Drug: Standard care +itraconazole 200mg

INTERVENTIONS:
Drug: Standard care +itraconazole 200mg — Is an antifungal used to treat a variety of fungal infections. It belongs to a class of drugs known as azole antifungals.
  Arms: Interventional arm
Drug: Chemotherapy — Standard Care (in control arm)
  Arms: Control arm

SUMMARY:
A prospective, randomized, controlled, parallel clinical trial will be conducted at Clinical Oncology and Nuclear Medicine Center at Mansoura University Hospital to assess the efficacy of Itraconazole as an adjuvant therapy in treatment of patients with acute myeloid Leukemia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Acute Myeloid leukemia, and aged 18 years or older
2. Patients whose ECOG performance status ranged from 0-2 and are fit for all treatments protocols

Exclusion Criteria:

1. Patients with any other types of malignancies rather than Leukemia and patients.
2. Patients with history alcohol intake, acute or chronic.
3. Patients with documented hypersensitivity or allergy to Itraconazole.
4. Patients suffer from chronic heart failure
5. Patients present with severe dehydration.
6. Patients with severe kidney dysfunction

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of blasts in bone marrow at d21 after induction | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed el-Husseiny shams, Principal Investigator — Professor Department of Clinical pharmacy and Pharmacy practice, Faculty of Pharmacy, Mansoura University; Moetaza Mahmoud Hassab Soliman, Study Director — Associate professor of Clinical Pharmacy, Clinical Pharmacy and Pharmacy Practice Department, Faculty of Pharmacy, Mansoura University; Noha Osama Mansour Mansour, Study Director — Lecturer of Clinical Pharmacy, Clinical Pharmacy and Pharmacy Practice Department, Faculty of Pharmacy, Mansoura University; Sara Mohamed Ali Atwa, Study Director — Lecturer of Medical Oncology, Department of Internal Medicine, Faculty of Medicine, Mansoura University
Locations (1):
- Clinical Oncology and Nuclear Medicine of Mansoura University Hospital, Mansoura,, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided